CLINICAL TRIAL: NCT06957470
Title: Comparison of the Effects in Target-controlled and Manually Controlled Total Intravenous Anesthesia on Postoperative Recovery and Patient Quality of Recovery in Septorhinoplasty Surgeries
Brief Title: TCI vs. Manuel TIVA in Septorhinoplasty Surgeries
Status: Active, not recruiting | Type: Observational
Sponsor: Bulent Ecevit University (Other)
Responsible Party: Principal Investigator, Büşra Sena Kuyumcu Hızal, medical doctor, Bulent Ecevit University
Other Study IDs: ZBEU-BHIZAL-001
Record Dates: First submitted 2025-03-29; First posted 2025-05-04 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Anesthesia
Keywords: septorhinoplasty; TIVA (total intravenous anesthesia); TCI (target controlled infusion)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- TCI (target controlled infusion): Patients in the TCI group will be anesthetized using the infusion method that selects the target area of effect of propofol and remifentanil.
  Interventions: Procedure: Total Intravenous Anesthesia
- MCI (manuel controlled infusion): Patients in the MCI group will be administered propofol and remifentanil as an infusion based on the anesthesiologist's observations.
  Interventions: Procedure: Total Intravenous Anesthesia

INTERVENTIONS:
Procedure: Total Intravenous Anesthesia — It is a general anesthesia technique performed through a combination of intravenous agents administered intravenously by various methods.

SUMMARY:
Septorhinoplasty is a surgical technique that can be used to correct various nasal deformities.Total intravenous anesthesia (TIVA) is a frequently preferred method as an anesthesia technique in septorhinoplasty surgeries.It has been reported that TIVA reduces the incidence of postoperative nausea and vomiting, is more successful in acute postoperative pain control compared to inhalational anesthesia, provides more stable hemodynamics, provides quicker awakening after anesthesia, is more effective in preventing recovery agitation and cough, and is effective in controlled hypotension.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-65 years with American Society of Anesthesiology (ASA) physical status I-II who will undergo Septorhinoplasty Surgery under general anesthesia will be included in the study.

Exclusion Criteria:

Patients who do not agree to participate in the study Patients under 18 and over 65 Patients with ASA score III and above Clinical diagnosis of neuropsychiatric disorders Those with a history of chronic NSAID, tranquilizer, opioid or sleeping pill use Clinical diagnosis of Serious cardiac diseases Clinical diagnosis of central-autonomic nervous system disease Clinical diagnosis of Coagulopathy Those with soybean oil allergy and a history of allergy to any study drug BMI >30 kg m2, pregnancy breastfeeding patients

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients aged 18-65 years with American Society of Anesthesiology (ASA) physical status I-II who will undergo Septorhinoplasty Surgery under general anesthesia
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
postoperative recovery | at postoperative 6 hours and 24 hours
  Postoperative recovery will evaluate with quality of recovery-40 questionnaire. quality of recovery-40 scores range from 40 (extremely poor quality of recovery) to 200 (excellent quality of recovery).
agitation during emergence | Postoperative 0 and 15. Minutes at the recovery room
  Agitation will evaluate with richmond sedation agitation scale. The richmond sedation agitation scale is a 10-point scale ranging from -5 to +4. Levels -1 to -5 denote 5 levels of sedation, starting with "awakens to voice" and ending with "unarousable." Levels +1 to +4 describe increasing levels of agitation.

SECONDARY OUTCOMES:
surgeon satisfaction | at the end of surgery
  5-point Likert Scale
postoperative pain | at the end of the surgery
  Numeric Rating Scale at the PACU
nausea and vomiting | Postoperative 0 hours at recovery room
  4-point Likert Scale

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Zonguladk Bulent ecevit University, Zonguldak, Kozlu
  - Bulent Ecevit University, Zonguldak, Zonguldak Province

IPD SHARING:
Plan to Share IPD: No